CLINICAL TRIAL: NCT02508441
Title: A Phase 1 Open-label First-in-human Dose-escalating Safety and Tolerability Study Evaluating Subcutaneous Administration of Andes-1537 for Injection in Patients With Advanced Unresectable Solid Tumors That Are Refractory to Standard Therapy or For Which No Standard Therapy is Available
Brief Title: Phase 1 Safety and Tolerability Study of Andes-1537 for Injection in Patients With Advanced Unresectable Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part 1 of the study was completed and the maximum tolerated dose determined. Part 2 of the study was terminated and will be conducted under a new protocol.
Sponsor: Andes Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB1537-001
Record Dates: First submitted 2015-07-15; First posted 2015-07-27 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Advanced Unresectable Solid Tumors
Keywords: Neoplasms; Solid Tumors; Advanced Malignancy; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Andes-1537 for Injection (Experimental): Part 1 is an open-label, dose-escalation study. Part 2 is an open-label, dose-expansion study.
  Interventions: Drug: Andes-1537 for Injection

INTERVENTIONS:
Drug: Andes-1537 for Injection — Part 1: Andes-1537 subcutaneous injection, 100 to 1000 mg twice a week per 4-week cycle
  Part 2: Andes-1537 subcutaneous injection, recommended phase 2 dose administered twice a week per 4-week cycle

SUMMARY:
This is a first-in-human, open-label, dose escalation and expansion, 2-part study to determine the safety, tolerability, and maximum tolerated dose of Andes-1537 for Injection in patients with advanced unresectable solid tumors that are refractory to standard therapy or for which no standard therapy is available.

DETAILED DESCRIPTION:
Part 1 is a dose-escalation study to establish the maximum tolerated dose based on dose-limiting toxicities and to evaluate the safety and tolerability of multiple doses of Andes-1537 for Injection in patients with advanced unresectable solid tumors that are refractory to standard therapy or for which no standard therapy is available. Part 2 is an open-label, dose-expansion study to determine the safety, tolerability, and preliminary efficacy of Andes-1537 in patients with advanced solid tumors. In part 2, patients will be enrolled and receive the recommended phase 2 dose established in part 1 based on the safety, tolerability, pharmacokinetics, and preliminary efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older
* Can understand and voluntarily sign an informed consent form prior to any study-related assessments or procedures, and are able to adhere to the study visit schedule and other protocol requirements
* Patient with documented pathological evidence of a cancer from which has developed advanced unresectable solid tumors that are, in the opinion of their treating physician, refractory to standard therapy or for which no standard therapy is available
* Consent to tumor biopsy from accessible tissue (optional in Part 1 and mandatory in Part 2)
* Have measureable disease by RECIST
* Have Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Have adequate organ function, confirmed by the following laboratory values obtained ≤ 3 days prior to the first treatment: absolute neutrophil count ≥ 1.5 × 10^9/L; hemoglobin ≥ 9 g/dL; platelets ≥ 100 × 10^9/L; aspartate transaminase and alanine transaminase ≤ 2.5 × upper limit of normal (ULN); serum total bilirubin ≤ 2.0 × ULN; serum creatinine ≤ 1.5 × ULN, or estimated or measured creatinine clearance ≥ 60 mL/min; prothrombin time, activated partial thromboplastin time ≤ 1.5 × ULN if not on anticoagulation therapy
* Female patients of childbearing potential must have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug.
* Male patients at screening must agree to practice adequate contraception from study entry through at least 6 months after discontinuation of study drug.

Exclusion Criteria:

* Have symptomatic central nervous system metastases. Patients with brain metastases that have been previously treated and are stable for ≥ 4 weeks or treated with gamma knife surgery and are stable for ≥ 2 weeks are allowed to enter the study.
* Have unstable angina, clinically significant cardiac arrhythmia, New York Heart Association Class 3 or 4 congestive heart failure, or prolonged QT interval corrected wave of greater than 470 ms.
* Receiving treatment with any medication known to produce QT prolongation within 7 days of study entry
* Have had prior systemic chemotherapy treatments or investigational modalities ≤ 5 half-lives or 4 weeks, whichever is shorter, prior to starting treatment with Andes-1537 or who have not recovered from side effects, grade 2 or greater, of such therapy (except alopecia)
* Have had major surgery ≤ 2 weeks prior to starting treatment with Andes-1537 or who have not recovered from side effects of such surgery
* Are pregnant or breastfeeding
* Have had DVT or venous thromboembolism within 6 weeks of study entry
* Have active uncontrolled bleeding or a known bleeding disorder
* Have any serious or unstable concomitant systemic conditions that are incompatible with this clinical study, including but not limited to substance abuse, psychiatric disturbance, or uncontrolled intercurrent illness (including active infection), arterial thrombosis, or symptomatic pulmonary embolism
* Have a known sensitivity to any of the components of Andes-1537
* Are unable or unwilling to follow protocol instructions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | First 4-week treatment cycle
  Determine maximum tolerated dose

SECONDARY OUTCOMES:
Adverse events | Safety evaluations will be measured through 28 days after last dose of Andes-1537
  Incidence of treatment-emergent adverse events
Safety laboratory tests | Safety evaluations will be measured through 28 days after last dose of Andes-1537
  Changes in baseline safety laboratory tests
Physical examinations | Safety evaluations will be measured through 28 days after last dose of Andes-1537
  Changes in baseline physical examination
Vital signs | Safety evaluations will be measured through 28 days after last dose of Andes-1537
  Changes in baseline vital signs
12-lead electrocardiogram (ECG) | First 4-week treatment cycle
  Changes in baseline ECG
Injection site reactions | Safety evaluations will be measured through 28 days after last dose of Andes-1537
  Incidence of injection site reactions
Pharmacokinetic parameters in Andes-1537 in blood and urine for single-dose and multiple-dose evaluation | Pre-treatment, following first dose and last dose of cycle 1 (4-week cycle), first dose of each additional cycle through study completion, and last visit
  Measure maximum concentration, time to maximum concentration, area under the curve, clearance, volume of distribution, and half-life
Pharmacodynamic parameters in blood and biopsy samples from accessible tissue | Pre-treatment and at 4 and 8 weeks for biopsy; blood samples at pre-treatment, every 8 weeks, and last visit
  Evaluate biomarkers in tissue and blood
Objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) with CT or MRI scan | Every 8 weeks following completion of 2 treatment cycles to cover from date of initiation until date of first documented progression or toxicity to Andes-1537, which ever comes first
  Changes in tumor size from baseline measurements

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Mount Zion, Helen Diller Family Comprehensive Cancer Center, Early Phase Clinical Trials, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No